CLINICAL TRIAL: NCT01570608
Title: Comparison of Ranibizumab (Lucentis) Monotherapy Versus Combination of Ranibizumab (Lucentis) With Photodynamic Therapy (Verteporfin) in Patients With Subfoveal Choroidal Neovascularisation Due to Age-Related Macular Degeneration - a Pilot Study
Brief Title: Lucentis KAV Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Ludwig Boltzmann Institute of Retinology and Biomicroscopic Laser Surgery (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EK 06-233-0107; 2006-006760-28 (EudraCT Number)
Record Dates: First submitted 2012-04-01; First posted 2012-04-04 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Age Related Macular Degeneration
Keywords: Ranibizumab; Bevacizumab; Verteporfin; age-related macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab; Verteporfin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- monotherapy arm (Active Comparator): patients receiving 3 initial Ranibizumab injections, thereafter as needed
  Interventions: Drug: Ranibizumab
- combined treatment arm (Active Comparator)
  Interventions: Drug: Ranibizumab; Drug: Verteporfin

INTERVENTIONS:
Drug: Ranibizumab — intravitreal injection 3 monthly injections thereafter as needed
Drug: Verteporfin — Verteporfin photodynamic therapy standard fluence
  Arms: combined treatment arm

SUMMARY:
Ranibizumab has been proven to be effective in large multicentre studies. However, the injections have to be repeated monthly. A combined therapy with the established photodynamic therapy might even be more effective, less intravitreal injections might be necessary due to a synergistic effect.

The study will be conducted to explore whether intravitreal ranibizumab in monotherapy or in combination with verteporfin photodynamic therapy under a new time regime is an effective, safe and convenient treatment for patients with subfoveal Choroidal Neovascularisation (CNV) secondary to Age-Related Macular Degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

* BCVA letter score in the study eye between 73-24 (approximately 20/40 to 20/320) using an ETDRS chart measured at 4 meters or Snellen equivalent
* CNV lesion of any type in the study eye which meets all the following characteristics as determined by fluorescein angiography:

  * Evidence that CNV extends under the geometric center of the foveal avascular zone.
  * The area of the CNV must occupy at least 50% of the total lesion.
  * The lesion must be ≤ 5400 microns in greatest linear dimension (GLD)
* For occult with no classic CNV, additionally recent disease progression as assessed by the Investigator is required defined as having at least one of the following criteria:

  * Blood associated with the lesion at baseline
  * Loss of VA in the previous 3 months defined as either ≥ 5 letters (ETDRS equivalent) as determined by protocol refraction and protocol measurements, or 2 or more lines using a Snellen or equivalent chart by standard examinations. ≥ 10% increase in the greatest diameter of the lesion in the previous 3 months as assessed by fluorescein angiography
* Willing to return for scheduled visits for a 12 month period
* Only one eye will be assessed in the study. If both eyes are eligible, the one with the worse visual acuity will be selected for treatment and study unless, based on medical reasons, the investigator deems the other eye the more appropriate candidate for treatment and study

Exclusion Criteria:

* Patients who have a BCVA of < 33 letters (approximately 20/200) in both eyes
* Prior treatment in the study eye with verteporfin, external-beam radiation therapy, vitrectomy, submacular surgery, other surgical intervention for AMD, or transpupillary thermotherapy
* Previous or current intravitreal drug delivery (e.g., intravitreal corticosteroid injection or device implantation) in the study eye
* Focal laser photocoagulation (juxta-, extra- or subfoveal) in the study eye
* Concomitant use of chronic NSAIDs or steroids (by any route) for the duration of study participation (chronic use is defined as multiple doses taken daily for three or more consecutive days at any time during the study). Note that ASA (aspirin) taken as "low dose" up to 100 mg qd for prophylaxis of MI and/or stroke is permitted during study
* Current use or of likely need for systemic medications known to be toxic to the lens, retina or optic nerve, including Deferoxamine, Chloroquine/ hydroxychloroquine (Plaquenil), Tamoxifen, Phenothiazines and Ethambutol is excluded
* History of glaucoma filtration surgery, corneal transplant surgery or extracapsular extraction of cataract with phacoemulsification within six months preceding Day One, or a history of post-operative complications within the last 12 months preceding Day One in the study eye (uveitis, cyclitis etc.)
* History of uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥ 25 mmHg despite treatment with topical anti-glaucomatous mediation).
* Aphakia or absence of the posterior capsule in the study eye
* Previous violation of the posterior capsule in the study eye is also excluded unless it occurred as a result of YAG posterior capsulotomy in association with prior, posterior chamber intraocular lens implantation
* Spherical equivalent of the refractive error in the study eye demonstrating more than -8 diopters of myopia
* Presence of a retinal pigment epithelial tear involving the macula in the study eye
* Angioid streaks or precursors of CNV in either eye due to other causes, such as ocular histoplasmosis, trauma, or pathologic myopia
* Active intraocular inflammation (grade trace or above) in the study eye
* Any active infection involving an eyeball adnexa
* Vitreous hemorrhage or history of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
number of injections | baseline-month 12
  Comparision of the number of required retreatments between the groups

SECONDARY OUTCOMES:
number of AE, SAE | 12 months
  number of AE and SAE
central retinal thickness | baseline-month 12
  central retinal thickness measured by OCT
distance acuity | baseline-month 12
  change of disance acuity measured by ETDRS letter scores

CONTACTS AND LOCATIONS:
Overall Officials: Ilse Krebs, MD, Study Director — Ludwig Boltzmann Institute for retinology and biomicroscopic Lasersurgery
Locations (3):
- Austria (3):
  - Department of OPhthalmology Medical center east, Vienna, Vienna
  - Department of Ophthalmology Rudolf foundation Clinic, Vienna, Vienna
  - Department of Ophthalmology, Hospital Hietzing, Vienna, Vienna